CLINICAL TRIAL: NCT03747419
Title: A Phase 2 Study of Avelumab in Combination With Bladder-Directed Radiation in Cisplatin-Ineligible Patients With Muscle-Invasive Urothelial Carcinoma of the Bladder
Brief Title: Avelumab and Radiation in Muscle-Invasive Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In agreement with the drug sponsor and the institution, the trial has been terminated due to slow accrual.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Kent Mouw, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-464
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer; Muscle Invasive Bladder Cancer
Keywords: Bladder Cancer; Bladder Carcinoma; Carcinoma of Bladder; Carcinoma of the Bladder; MIBC; Muscle Invasive Bladder Cancer; Muscle-Invasive Urothelial Carcinoma of the Bladder; Immunotherapy; Avelumab; Radiation and Immunotherapy; No cisplatin; Cisplatin Ineligible; Cisplatin-Ineligible; T2 Disease; T3 Disease; T4 Disease; squamous bladder cancer; adenocarcinoma bladder cancer; micropapillary bladder cancer; Inability to receive cisplatin-based chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — avelumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab and Bladder-Directed Radiation (Experimental): * Avelumab will be administered every 2 weeks intravenously for 6 doses unless there is unacceptable toxicity
  * Two radiation dose regimens are allowed, and the regimen selected is at the discretion of the treating radiation oncologist
  Interventions: Drug: Avelumab; Radiation: Radiation

INTERVENTIONS:
Drug: Avelumab — Avelumab is a form of immunotherapy, which means it is designed to help the patient's immune system kill cancer cells.
  Other Names: Bavencio
Radiation: Radiation — Cancer treatment that uses ionizing radiation to kill cancer cells.

SUMMARY:
This research study is studying the effects of adding a certain type of immunotherapy to standard bladder-directed radiation as a treatment for muscle-invasive urothelial carcinoma of the bladder.

The drug in this study is: Avelumab (also known as BAVENCIO®)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved the use of avelumab and bladder-directed radiation together for this specific disease but avelumab has been approved for other uses.

While bladder-directed radiation is a standard treatment option for muscle-invasive urothelial carcinoma of the bladder, the use of avelumab in combination with bladder radiation in patients with urothelial carcinoma of the bladder is investigational. Radiation is used in the treatment of muscle-invasive bladder cancer, and avelumab has been approved by the FDA in patients with more advanced stages of this disease. Avelumab is a form of immunotherapy, which means it is designed to help the immune system fight cancer cells together with standard cancer treatments like radiation. Avelumab is currently approved by the FDA for the treatment of metastatic Merckel cell carcinoma (mMCC) and platinum-refractory metastatic urothelial carcinoma.

The purpose of this study is to test whether the combination of immunotherapy and bladder directed radiation is effective in treating muscle-invasive bladder cancer. The study will also measure other outcomes such as participant's overall health and quality of life during and after treatment. In addition, the investigators will determine if certain biomarkers are correlated with outcomes following treatment with immunotherapy and radiation.

ELIGIBILITY:
Subjects must meet all of the following applicable inclusion criteria to participate in the study.

Inclusion Criteria:

* Histologically confirmed transitional cell (urothelial) carcinoma of the bladder that is invasive into the muscularis propria (≥T2 disease) within 6 months of enrollment date. The presence of variant histologies (squamous, adenocarcinoma, micropapillary, etc.) is allowed. Note: A prior diagnosis of non-muscle-invasive bladder cancer (≤T1) managed with transurethral resection with or without intravesicular therapy (now with muscle invasion) is allowed.
* Inability to receive cisplatin-based chemotherapy, as defined by creatinine clearance <60 ml/min, ECOG PS ≤2, grade 2 or higher hearing loss, NYHA class 3 or higher, neuropathy (grade 2 or higher), or patient refusal to receive cisplatin-based chemotherapy.

Additional Inclusion Criteria:

* Male or female subjects aged ≥18 years
* ECOG performance status ≤2 or Karnofsky score ≥60% (see Appendix A)
* Life expectancy of greater than 1 year
* Demonstrate normal organ and marrow function
* Estimated creatinine clearance > 30 mL/min according to the Cockcroft-Gault formula.
* Women of child-bearing age must have a negative serum pregnancy test at screening.
* Women of child-bearing potential and men must agree to use a highly effective method of contraception (hormonal or barrier method of birth control, or abstinence) beginning prior to study entry, for the duration of study participation, and for at least 30 days after last avelumab treatment administration if the risk of conception exists
* Ability to start study treatment (first cycle of Avelumab) within 1-8 weeks of the most recent pre-study TURBT.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Prior intravenous therapy for treatment of bladder cancer
* Prior pelvic radiation
* Any component of small cell histology in the bladder biopsy
* Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroid, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) are allowed.
* History of another malignancy within 5 years prior to randomization except for: non-muscle-invasive bladder cancer (i.e., ≤T1), completely resected basal cell or squamous cell skin cancer, completed resected carcinoma-in-situ of any site, or localized prostate cancer managed definitively with a non-radiation based approach.

Additional Exclusion Criteria:

* Evidence of lymph node involvement or metastatic disease on CT of the chest, abdomen, and pelvis. To be considered positive, a lymph node must measure >15 mm in short axis.
* Clinically significant (i.e. active) cardiovascular disease: symptomatic congestive heart failure (≥ New York Heart Association Classification Class II), unstable angina pectoris, serious cardiac arrhythmia requiring medication, or CVA/stroke/MI (< 6 months prior to enrollment)
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
* Breast feeding women who are unwilling to stop breastfeeding during treatment and for at least one month after the duration of treatment
* Patients with known history of testing positive for HIV or known acquired immunodeficiency syndrome
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Active infection requiring intravenous antibiotic therapy
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines
* Major surgery within the last 30 days (with the exception of TURBT).
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* Prior organ transplantation including allogenic stem-cell transplantation
* Patient is unwilling to stop (or wishes to start) taking herbal and natural remedies that may have immune-modulating effects during the study period
* Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Pregnant women are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Mouw, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 patients were enrolled out of 17 that consented to the study. The target enrollment was 24 patients prior to study closure due to slow accrual.
Pre-assignment Details: Patients must have muscle invasive (T2-T4a) urothelial bladder carcinoma. They must also not be eligible for cisplatin-based chemotherapy.
Period: Overall Study
Arm/Group | Avelumab and Bladder-Directed Radiation
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 14 patients with muscle-invasive (T2-T4a) urothelial bladder carcinoma, not eligible for cisplatin-based chemotherapy
Arm/Group | Avelumab and Bladder-Directed Radiation
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status scores were assessed by treating physician within 28 days prior to registration. Higher score means worse outcome at baseline:
  0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. = Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    ECOG = 0 | 5
    ECOG = 1 | 5
    ECOG = 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Clinical Response Rate
Description: Measured by the complete clinical response rate at 3 months following completion of radiation, followed by every 3 months until 2 years after registration, then every 6 months up to a maximum of 3 years after registration. Clinical response is assessed by cystoscopy, urine cytology, and CT Chest/Abdomen/Pelvis. No evidence of disease on these assessments at a given time point suggests a Complete Clinical Response at that time point.
Time Frame: 3 months following completion of radiation; then every 3 months until 2 years after registration; then every 6 months up to a maximum of 3 years after registration
Population: 2 participants withdrew consent prior to completing protocol therapy and therefore could not be evaluated for the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab and Bladder-Directed Radiation
Number analyzed (Participants) | 12
Participants
  Subjects that reached Complete CR at 3 months following completion of radiation | 5
  Subjects that never reached Complete CR during FU | 3
  Subjects that reached Complete CR during FU but after 3 months following completion of radiation | 4

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS)
Time Frame: 3 years
Population: 2 participants withdrew consent prior to completing protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab and Bladder-Directed Radiation
Number analyzed (Participants) | 12
Participants
  Deaths due to progressive disease during FU | 5
  Deaths due to unrelated condition during FU | 2
  Subjects alive at time of study closure | 4
  Subjects alive at time of study withdrawal during FU | 1

3. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) as assessed by imaging, cystoscopy, and cytology.
Time Frame: 3 years
Population: 2 participants withdrew consent prior to completing protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab and Bladder-Directed Radiation
Number analyzed (Participants) | 12
Participants
  Disease progression after treatment | 5
  No disease progression after treatment | 7

4. Secondary Outcome: Metastases-free Survival
Description: Metastases-free survival (MFS) as assessed by imaging.
Time Frame: 3 years
Population: 2 participants withdrew consent prior to completing protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab and Bladder-Directed Radiation
Number analyzed (Participants) | 12
Participants
  Metastases after treatment | 5
  No metastases after treatment | 7

5. Secondary Outcome: Locoregional Recurrence Rate
Description: Locoregional recurrence rate (LRR) as assessed by imaging.
Time Frame: 3 years
Population: 2 participants withdrew consent prior to completing protocol therapy, and 1 participant withdrew consent during FU. Therefore, they could not be evaluated for overall survival.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab and Bladder-Directed Radiation
Number analyzed (Participants) | 12
Participants
  Locoregional recurrence after treatment | 1
  No locoregional recurrence after treatment | 11

6. Secondary Outcome: Change in Quality of Life Outcomes
Description: Quality of Life Outcomes (QoL) as measured by patient report on questionnaires. Patients are given a statement and must assign a number to assess how the statement applies to them in the past 7 days. 0=Not at all; 1=A little bit; 2=Somewhat; 3=Quite a bit; 4=Very much. QoLs were collected at baseline, end of radiation, 3 months post-radiation completion, then every 3 months through year 2 after treatment.
  Median scores and interquartile ranges were calculated for baseline, 3 months post-radiation completion, and 2 years post-treatment. 3 months post-RT was selected to coincide with the primary outcome timeframe. Year 2 was selected due to the number of patients that reached this point during follow up; most patients did not surpass year 2.
  Higher score means worse outcome for questions regarding diarrhea, urinary frequency & burning, and being bothered by treatment. Higher score means better outcome for questions regarding being content with quality of life and control over bowels.
Time Frame: Baseline; 3 months following completion of radiation; 2 years after treatment
Population: One participant declined to complete QoL forms during treatment and follow up.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Avelumab and Bladder-Directed Radiation
Number analyzed (Participants) | 13
score on a scale
  Baseline Median Score "I am bothered by side effects of treatment" | 0 [0 to 0]
  Baseline Median Score "I am content with the quality of my life right now" | 2 [2 to 3]
  Baseline Median Score "I have control of my bowels" | 3 [2 to 4]
  Baseline Median Score "I urinate more frequently than usual" | 2.5 [1.75 to 3.25]
  Basline Median Score "I have diarrhea" | 0 [0 to 0]
  Baseline Median Score "It burns when I urinate" | 0 [0 to 1]
  3 months post-RT Median Score "I am bothered by side effects of treatment" | 0 [0 to 0]
  3 months post-RT "I am content with the quality of my life right now" | 3 [2 to 3]
  3 months post-RT Median Score "I have control of my bowels" | 1.5 [1.25 to 3]
  3 months post-RT Median Score "I urinate more frequently than usual" | 2 [1.8125 to 2.875]
  3 months post-RT Median Score "I have diarrhea" | 0.5 [0 to 1.75]
  3 months post-RT Median Score "It burns when I urinate" | 0 [0 to 0]
  2 Year Median Score "I am bothered by side effects of treatment" | 0 [0 to 0]
  2 Year Median Score "I am content with the quality of my life right now" | 3 [3 to 4]
  2 Year Median Score "I have control of my bowels" | 3 [1.3125 to 3]
  2 Year Median Score "I urinate more frequently than usual" | 0 [0 to 2.65625]
  2 Year Median Score "I have diarrhea" | 0 [0 to 1.4375]
  2 Year Median Score "It burns when I urinate" | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Baseline; every 2 weeks during Avelumab treatment; 30 post-completion of Avelumab treatment; 3 months post-completion of radiation; then every 3 months until 2 years post-treatment; then every 6 months during years 3-5 post-treatment
Description: Assessed by research nurses, medical oncologists, physician assistants, nurse practitioners
Arm/Group | Avelumab and Bladder-Directed Radiation
All-Cause Mortality (participants affected / at risk) | 7/14
Serious Adverse Events (participants affected / at risk) | 4/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab and Bladder-Directed Radiation (N=14)
Aspartate aminotransferase increased (Investigations) | 1 (1) — Grade 4, Unlikely related to Avelumab or Radiation
Alkaline phosphatase increased (Investigations) | 1 (1) — Grade 3, Unlikely related to RT and Avelumab
Creatinine increased (Investigations) | 1 (1) — Grade 3, unlikely related to RT
Fatigue (General disorders) | 1 (1) — Grade 3, Definitely related to RT, Possibly related to Avelumab
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Grade 3, Unlikely related to RT or Avelumab
Hypotension (Vascular disorders) | 1 (1) — Grade 2, Definitely related to RT, unlikely related to Avelumab
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) — Grade 3, Possibly related to RT, Unrelated to Avelumab
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — Grade 3, Probably related to RT, Unlikely related to Avelumab
Lung infection (Infections and infestations) | 1 (1) — Grade 3, Unrelated to RT and Avelumab
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab and Bladder-Directed Radiation (N=14)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 6 (6)
Fever (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 6 (6)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination was due to slow accrual. 14 out of 24 patients were accrued during the duration of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT03747419/Prot_SAP_000.pdf